CLINICAL TRIAL: NCT06022484
Title: How Many Days Will You Delay Before a MRI When You Have Low Back Pain?
Brief Title: Magnetic Resonance Imaging and Acute Low Back Pain
Status: Completed | Type: Observational
Sponsor: International Institute of Behavioral Medicines (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-005
Record Dates: First submitted 2023-08-21; First posted 2023-09-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Acute Low Back Pain
Keywords: Low back pain; Magnetic Resonance Imaging; Catastrophizing; Anxiety; Red flags
MeSH Terms: conditions — Low Back Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with acute low back pain: No intervention.
  Interventions: Other: The present study does not contain any intervention
- General practitioners who treat people with acute low back pain: No intervention.
  Interventions: Other: The present study does not contain any intervention

INTERVENTIONS:
Other: The present study does not contain any intervention — The present study does not contain any intervention

SUMMARY:
This is a behavioral observational study aimed at understanding the limit of tolerance (in days) of ideally performing a Magnetic Resonance Imaging (MRI) by people with acute low back pain. It consists of a short self-administered questionnaire. Relationships between low back pain intensity, maladaptive thoughts and awaited days before ideally requesting a MRI will be evaluated.

DETAILED DESCRIPTION:
This is a behavioral observational study aimed at understanding the limit of tolerance (in days) of ideally performing a Magnetic Resonance Imaging (MRI) by people with acute low back pain (LBP) and by general practitioners (GP).

Literature pointed out that LBP is a common occurrence in people, with high rates of self-resolution in the absence of red flags (i.e. possible indicators of serious spinal pathology).

In Italy there is an over-prescription of MRI despite international guidelines go the opposite way.

The study consists of a short self-administered questionnaire which will be given to people and GP to complete. In more details, the survey is made of 3 questions collecting information on the limit of tolerance (in days) before requesting (people) and prescribing (GP) a MRI for the lumbar tract of the spinal column.

Further, participants will have to complete a self-administered pain intensity numerical rating scale, along with catastrophizing and anxiety self-administered questionnaires.

Descriptive statistics will be presented by taking into account the socio-demographic characteristics of the sample being investigated. Statistical correlations between participants' answers and the scores from the questionnaires will be also evaluated.

This study investigates the relationships among acute low back pain, the intention of persons/GP to request/prescribe a MRI despite the absence of red flags, mood disorders and maladaptive thoughts.

ELIGIBILITY:
Inclusion Criteria:

* Having acute low back pain (i.e., a pain lasting no more than 6 weeks)
* Adult age
* Ability to understand the Italian language

Exclusion Criteria:

* Mental deficits
* Refuse to adhere to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult people with acute low back pain (i.e., a pain lasting no more than 6 weeks).
  General practitioners who are involved in the managment of people with acute low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Two questions on limit of tolerance | Up to the first day
  Design of questions which investigates the limit of tolerance of requesting and prescribing a MRI; score is expressed as "number of days" (neither min nor max values are stated a priori).

SECONDARY OUTCOMES:
NRS | Up to the first day
  pain intensity Numerical Rating Scale; score 0-10 with higher estimates indicating higher levels of pain intensity
PCS | Up to the first day
  Pain Catastrophizing Scale; score 0-52 with higher estimates indicating higher levels of catastrophizing.
ZUNG | Up to the first day
  Zung Self-Rating Anxiety Scale; score 20-80 with higher estimates indicating higher levels of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Rocca, Calosso, Italy

IPD SHARING:
Plan to Share IPD: No